CLINICAL TRIAL: NCT04532749
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of Seltorexant 20 mg as Adjunctive Therapy to Antidepressants in Adult and Elderly Patients With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant Therapy
Brief Title: A Study of Seltorexant as Adjunctive Therapy to Antidepressants in Adult and Elderly Participants With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 42847922MDD3002 was stopped based on the interim analysis (IA) results as recommended by the Independent Data Monitoring Committee (IDMC)
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108805; 42847922MDD3002 (Other: Janssen Research & Development, LLC); 2020-000338-16 (EudraCT Number)
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seltorexant (Experimental): Participants will receive Seltorexant orally once daily from Day 1 to Day 42 (until the end of Week 6).
  Interventions: Drug: Seltorexant
- Placebo (Placebo Comparator): Participants will receive matching placebo tablets orally once daily from Day 1 to Day 42 (until the end of Week 6).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seltorexant — Participants will receive Seltorexant tablets.
  Arms: Seltorexant
Drug: Placebo — Participants will receive matching placebo tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Seltorexant compared with placebo as adjunctive therapy to an antidepressant in improving depressive symptoms in participants with major depressive disorder with insomnia symptoms (MDDIS) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common, serious, recurrent disorder. Seltorexant (JNJ-42847922) is a potent and selective antagonist of the human orexin-2 receptor (OX2R) that is being developed for the adjunctive treatment of MDDIS. The hypothesis for this study is that adjunctive treatment with seltorexant is superior to placebo in treating depressive symptoms, as measured by change in Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to Day 43 in adult and elderly participants with MDDIS who have had an inadequate response to treatment with a SSRI/SNRI. The study will be conducted in 3 phases: a screening phase (up to 30 days), a double-blind (DB) treatment phase (43 days), and a post treatment follow-up phase (7 to 14 days after DB treatment phase). Total duration of study is up to 12 weeks. Efficacy, safety, pharmacokinetics, and biomarkers will be assessed at specified time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic and statistical manual of mental disorders-5th edition (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 Axis I disorders-clinical trials version (SCID-CT) diagnosed with first depressive episode prior to age 60. The duration of the current depressive episode must be less than or equal to (<=) 24 months
* Have had an inadequate response to at least 1 but no more than 2 antidepressants, administered at an adequate dose and duration in the current episode of depression. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression. An inadequate response is defined as less than (<) 50 percent (%) reduction but with some improvement (that is, improvement greater than [>] 0%) in depressive symptom severity with residual symptoms other than insomnia present, and overall good tolerability, as assessed by the MGH-ATRQ
* Is receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any formulation and available in the participating country: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at therapeutic dose level) for at least 6 weeks, and for no greater than 18 months in the current episode
* Have a hamilton depression rating scale (HDRS)-17 total score greater than or equal to (>=) 20 at the first screening interview, must not demonstrate a clinically significant improvement (that is [ie], an improvement of > 20 % on their HDRS-17 total score) from the first to the second independent HDRS-17 rating, and must have a HDRS-17 total score >= 18 at the second screening interview
* Have a patient version of the Insomnia Severity Index (ISI) total score >=15 as well as a clinician version of the ISI total score >=15 at the second screening visit
* Body mass index (BMI) between 18 and 40 kilogram per meter square (kg/m^2) inclusive (BMI=weight/height^2)
* Participant must be medically stable on the basis of clinical laboratory tests performed at screening
* Participant must be medically stable on the basis of the following: physical examination (including a brief neurological examination), vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed at screening and baseline

Exclusion Criteria:

* Has a recent (last 3 months) history of, or current signs and symptoms of, severe renal insufficiency (creatinine clearance [CrCl] < 30 milliliter per minute [mL/min]); clinically significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic or endocrine disorders and uncontrolled Type 1 or Type 2 diabetes mellitus
* Has clinically significant hepatic disease as defined by >=2*Upper Limit of Normal (ULN) increase of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at screening
* Has a history of treatment-resistant MDD, defined as a lack of response to 2 or more adequate antidepressant treatments in the current episode, as indicated by no or minimal (< 25% improvement in symptoms) when treated with an antidepressant of adequate dose (per massachusetts general hospital-antidepressant treatment response questionnaire [MGH-ATRQ]) and duration (at least 6 weeks).
* Has history or current diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, or somatoform disorders
* Has any significant primary sleep disorder, including but not limited to obstructive sleep apnea, restless leg syndrome, or parasomnias. Participants with insomnia disorder are allowed
* Has a history of moderate to severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (80):
- United States (26):
  - Altea Research Institute, Phoenix, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Behavioral Research Specialists LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Alliance for Research, Long Beach, California
  - Excell Research Inc, Oceanside, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Pharmax Research Clinic Inc, Miami, Florida
  - Innova Clinical Trials, Miami, Florida
  - Harmony Clinical Research Inc, North Miami Beach, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Synexus Research Orlando, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Compass Research LLC-Bioclinica Research, The Villages, Florida
  - Synexus Clinical Research US Inc, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Michigan Clinical Research Institute, Ann Arbor, Michigan
  - Eastside Comprehensive Medical Services, New York, New York
  - Community Research Management Associates, Inc., Cincinnati, Ohio
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - Intend Research, Norman, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - InSite Clinical Research LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
- Argentina (10):
  - Clínica Privada Banfield S.A, Banfield
  - STAT Research S A, Buenos Aires
  - NOVAIN Neurociencias Group, Buenos Aires
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Sanatorio Prof. Leon S. Morra, Córdoba
  - INSA Instituto de Neurociencias San Agustín, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Chile (4):
  - Psicomed Estudios Medicos, Antofagasta
  - BioMedica Research Group, Santiago
  - CeCim - Centro de Estudios Clinicos e Investigacion Medica, Santiago
  - Hospital Dr Hernan Henriquez Aravena, Temuco
- Denmark (2):
  - Ålborg Universitetshospital, Aalborg
  - Psykiatrisk Center Nordsjaelland, Hillerød
- Finland (5):
  - Eira Hospital, Helsinki
  - Mederon LTD at ARTES, Helsinki
  - Savon Psykiatripalvelu, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu, Rauma
- Malaysia (4):
  - Hospital Kuala Lumpur, Jalan Pahang
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Sibu, Sibu
  - Sunway Medical Centre, Sunway City
- Poland (6):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - Synexus Polska Sp z o o Oddzial w Katowicach, Katowice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Synexus Polska Sp z o o, Lodz
  - Centrum Medyczne Luxmed Sp z o o, Lublin
- Slovakia (4):
  - Psychiatricka Ambulancia Mentum S.R.O., Bratislava
  - Psychiatricka Ambulancia Centrum Zdravia R.B.K. S.R.O., Svidník
  - Crystal Comfort s.r.o., Vranov nad Topľou
  - BONA MEDIC, s.r.o., Zlaté Moravce
- South Korea (8):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Eulji General Hospital, Seoul
- Ukraine (11):
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - CNPE'Kherson Regional Institution of Mental Care'of Kherson Regional Council, Kherson
  - Cnce 'Kyiv City Psychoneurological Hospital #2' of Executive Body of Kyiv City Council (Kcsa), Kyiv
  - Main Military Clinical Hospital of MDU, Kyiv
  - Kyiv Clinical Railway Hospital #2 of the Branch Health Care Center of the PJSC Ukrainian Railway, Kyiv
  - CNCE of the Lviv Regional Council 'Lviv Regional Clinical Psychiatric Hospital', Lviv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - CNCE Odesa regional psychiatric hospital #2 Odesa regional council, Oleksandrivka
  - Poltava O.F. Maltsev RC Psychiatric Hospital Dept #9 (Ad-P Dept) HSEIU Ukrainian MSA, Poltava
  - CNCE 'Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council', Smila
  - CI O.I. Yuschenko VRPsH Depts #7 & #10 M.I. Pyrogov VNMU, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with major depressive disorder with insomnia symptoms (MDDIS) who had an inadequate response to an ongoing antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) were randomized in the study. Study consisted of screening phase, double-blind (DB) treatment phase and a post-treatment follow-up (FU) phase.
Groups:
- Seltorexant: During DB treatment phase, participants received seltorexant 20 milligrams (mg) tablet orally once daily from Day 1 to Day 42. Participants were then followed up for safety up to 7 to 14 days after end of DB treatment at Day 43 (up to Day 57) during the follow-up phase. Participants who discontinued study drug prior to Day 35 were encouraged to have additional follow-up visits every 2 weeks until Day 50 to 57.
- Placebo: During DB treatment phase, participants received placebo matching to seltorexant tablet orally once daily from Day 1 to Day 42. Participants were then followed up for safety up to 7 to 14 days after end of DB treatment at Day 43 (up to Day 57) during the follow-up phase. Participants who discontinued study drug prior to Day 35 were encouraged to have additional follow-up visits every 2 weeks until Day 50 to 57.
Period: DB Treatment Phase (Day 1 to Day 43)
Arm/Group | Seltorexant | Placebo
Started | 107 | 105
Completed | 101 | 89
Not Completed | 6 | 16
Not completed — Adverse Event | 1 | 6
Not completed — Lack of Efficacy | 2 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Other | 1 | 2
Period: Follow-up Phase (Day 44 to Day 57)
Arm/Group | Seltorexant | Placebo
Started | 103 (Included 3 participants (2 due to lack of efficacy + 1 due to other unspecified reason) who discontinued DB treatment phase but continued study and entered the follow-up phase. One participant completed DB treatment phase but was lost to follow-up for the study and thus did not enter follow-up phase.) | 98 (Included 9 participants (5 due to adverse events + 2 due to lack of efficacy + 1 due to protocol violation + 1 study termination by sponsor) who discontinued DB treatment phase but continued study and entered follow-up phase.)
Completed | 102 | 92
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Seltorexant: During DB treatment phase, participants received seltorexant 20 mg tablet orally once daily from Day 1 to Day 42. Participants were then followed up for safety up to 7 to 14 days after end of DB treatment at Day 43 (up to Day 57) during the follow-up phase. Participants who discontinued study drug prior to Day 35 were encouraged to have additional follow-up visits every 2 weeks until Day 50 to 57.
- Total: Total of all reporting groups
Arm/Group | Seltorexant | Placebo | Total
Number analyzed (Participants) | 107 | 105 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (13.87) | 48.8 (14.40) | 49.5 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 83 | 161
  Male | 29 | 22 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 33 | 71
  Not Hispanic or Latino | 68 | 72 | 140
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 14 | 23
  White | 90 | 87 | 177
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 13 | 14 | 27
  Chile | 3 | 4 | 7
  Denmark | 1 | 1 | 2
  Finland | 10 | 9 | 19
  Malaysia | 1 | 0 | 1
  Poland | 6 | 4 | 10
  Slovakia | 9 | 8 | 17
  Korea, South | 3 | 4 | 7
  Ukraine | 23 | 25 | 48
  United States | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 43 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS was a clinician-rated scale designed to measure depression severity and detected changes due to antidepressant treatment. The scale consisted of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score was the sum of scores from individual question items, which ranged from 0 to 60, higher scores represented a more severe condition. Negative change in MADRS total score indicated improvement.
Time Frame: Baseline (Day 1), Day 43
Population: The full analysis set 1 (FAS1) included all randomized participants who received at least 1 dose of study intervention in the DB phase and had baseline MADRS total score greater than or equal to (>=) 24 (per interactive web response system [IWRS]). Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 101 | 89
Units on a scale | -14.0 (10.46) | -13.1 (9.51)
Statistical Analysis 1: Comparison: Seltorexant vs Placebo; Test type: Superiority; p = 0.411, Mixed Model Repeated Measures (MMRM); Least square (LS) mean difference = -1.2, 95% CI 2-sided [-4.00 to 1.64], Standard Error of Mean 1.43

2. Secondary Outcome: Change From Baseline to Day 43 in the MADRS Without Sleep Item (MADRS-WOSI) Total Score
Description: The MADRS was a clinician-rated scale designed to measure depression severity and detected changes due to antidepressant treatment. MADRS-WOSI was defined as the full MADRS without the sleep item. The MADRS-WOSI scale consisted of 9 items (apparent sadness, reported sadness, inner tension, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). Higher scores represented a more severe condition. MADRS-WOSI total score was the sum of scores from individual question items, which ranged from 0 to 54, higher scores represented a more severe condition. Negative change in MADRS total score indicated improvement.
Time Frame: Baseline (Day 1), Day 43
Population: FAS1 included all randomized participants who received at least 1 dose of study intervention in the DB phase and had baseline MADRS total score >=24 (per IWRS). Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 101 | 89
Units on a scale | -12.0 (9.27) | -11.3 (8.44)
Statistical Analysis 1: Comparison: Seltorexant vs Placebo; In accordance with protocol predefined testing sequence, statistical significance of the primary endpoint was required before testing the first secondary endpoint (MADRS-WOSI) and thus, a formal statistical testing was not performed; Test type: Superiority; p = 0.473, MMRM model; LS mean difference = -0.9, 95% CI 2-sided [-3.41 to 1.59], Standard Error of Mean 1.27

3. Secondary Outcome: Change From Baseline to Day 43 in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD; Short Form 8a) T-score
Description: PROMIS-SD Short Form 8a: static 8-item questionnaire, assessed self-perceptions of sleep initiation (2 items), quality of sleep (3 items), early morning feelings (2 items), worrying about sleep (1 item). Each question has 5 options ranged 1 to 5. The "direction" of responses was not same, sometimes "not at all" =more sleep disturbance; sometimes "not at all" =less sleep disturbance. Total raw score for short form with all questions answered was sum of values of response to each question, total score ranged 8 to 40. Lower scores=less sleep disturbance. Total raw score converted into T-score. T-score rescaled the raw score into standardized score with mean-50; SD-10. Negative changes in scores=improvement. Higher PROMIS T-score represents more concept measured. Negatively worded (like sleep disturbance), T-score of 60 was one SD worse than average. By comparison, T-score of 40 was one SD better than average. T-score of 50 or above was clinically significant level of sleep disturbance.
Time Frame: Baseline (Day 1), Day 43
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 101 | 89
T-score | -13.7 (11.06) | -11.9 (11.83)
Statistical Analysis 1: Comparison: Seltorexant vs Placebo; In accordance with protocol predefined testing sequence, statistical significance of the primary endpoint was required before testing the second secondary endpoint (PROMIS-SD; Short Form 8a) and thus, a formal statistical testing was not performed; Test type: Superiority; p = 0.167, MMRM Model; LS mean difference = -2, 95% CI 2-sided [-4.87 to 0.85], Standard Error of Mean 1.45

4. Secondary Outcome: Change From Baseline to Day 43 in the 6-item MADRS (MADRS-6) Total Score
Description: The 6-item MADRS was a clinician-administered scale designed to measure the core symptoms of depression severity and detected changes due to antidepressant intervention. It is a subset of MADRS (10-item). The MADRS-6 subscale score was the sum of scores for the following MADRS items: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts. Each item was scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms), the overall score ranges from 0 to 36, higher scores represented a more severe condition. Negative changes in MADRS-6 total score indicate improvement.
Time Frame: Baseline (Day 1), Day 43
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 101 | 89
Units on a scale | -9.1 (6.86) | -8.1 (6.37)

5. Secondary Outcome: Percentage of Participants Who Achieved Response on Depressive Symptoms Scale Based on MADRS Total Score at Day 43
Description: Percentage of participants who achieved response on depressive symptoms scale based on MADRS total score at Day 43 were reported. Responders were defined as participants with a >=50 percent (%) improvement in the MADRS total score from baseline to a given timepoint. The MADRS was a clinician-rated scale designed to measure depression severity and detected changes due to antidepressant treatment. The scale consisted of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score was the sum of scores from individual question items, which ranged from 0 to 60, higher scores represented a more severe condition. Negative change in MADRS total score indicated improvement.
Time Frame: At Day 43
Population: FAS1 included all randomized participants who received at least 1 dose of study intervention in the DB phase and had baseline MADRS total score >=24 (per IWRS).
Measure: Number; unit: Percentage of participants
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 105 | 102
Percentage of participants | 42.9 | 36.3

6. Secondary Outcome: Change From Baseline to Day 43 in Patient Health Questionnaire, 9-item (PHQ-9) Total Score
Description: The PHQ-9 was a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) major depressive disorder (MDD) criteria. Each item was rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses were summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 was categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). Negative changes in PHQ-9 total score indicated improvement.
Time Frame: Baseline (Day 1), Day 43
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Seltorexant | Placebo
Number analyzed (Participants) | 101 | 89
Units on a scale | -8.8 (6.44) | -8.1 (6.27)

ADVERSE EVENTS:
Time Frame: Double-blind (DB) Phase: From Day 1 up to Day 43; Follow up Phase: From Day 44 to Day 57
Description: DB Phase: The safety analysis set included all randomized participants who received at least 1 dose of study intervention in the DB phase. Follow-up Phase: The follow-up analysis set included all randomized participants who entered the follow up phase.
Groups:
- DB Phase: Seltorexant: During DB treatment phase, participants received seltorexant 20 mg tablet orally once daily from Day 1 to Day 42.
- DB Phase: Placebo: During DB treatment phase, participants received placebo matching to seltorexant tablet orally once daily from Day 1 to Day 42.
- Follow-up Phase: Seltorexant: Participants who received seltorexant 20 mg and completed DB treatment phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB treatment at Day 43 (up to Day 57). Participants who discontinued study drug prior to Day 35 were encouraged to have additional follow-up visits every 2 weeks until Day 50 to 57.
- Follow-up Phase: Placebo: Participants who received placebo and completed DB treatment phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB treatment at Day 43 (up to Day 57). Participants who discontinued study drug prior to Day 35 were encouraged to have additional follow-up visits every 2 weeks until Day 50 to 57.
Arm/Group | DB Phase: Seltorexant | DB Phase: Placebo | Follow-up Phase: Seltorexant | Follow-up Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/105 | 0/103 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/107 | 2/105 | 0/103 | 0/98
Other Adverse Events (participants affected / at risk) | 14/107 | 11/105 | 0/103 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Seltorexant (N=107) | DB Phase: Placebo (N=105) | Follow-up Phase: Seltorexant (N=103) | Follow-up Phase: Placebo (N=98)
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Seltorexant (N=107) | DB Phase: Placebo (N=105) | Follow-up Phase: Seltorexant (N=103) | Follow-up Phase: Placebo (N=98)
Headache (Nervous system disorders) | 14 | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will delay to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT04532749/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04532749/SAP_001.pdf